CLINICAL TRIAL: NCT06626737
Title: Dapagliflozin for Preventing Acute Graft-versus-Host Disease in Allogeneic Hematopoietic Cell Transplantation: A Prospective, Single-Arm Study
Brief Title: Dapagliflozin in Allo-HCT for aGVHD
Acronym: DAPALAG-01
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024348
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Graft-versus-host Disease (GVHD)
Keywords: Dapagliflozin; Graft-versus-host disease; Allogeneic hematopoietic cell transplantation
MeSH Terms: conditions — Graft vs Host Disease | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dapagliflozin arm (Experimental): Participants will take Dapagliflozin10mg every day in -1 to 14 days.
  Interventions: Drug: Dapagliflozin (DAPA)

INTERVENTIONS:
Drug: Dapagliflozin (DAPA) — Participants will take Dapagliflozin 10mg every day in -1 to 14 days

SUMMARY:
The goal of this clinical trial is to learn if Dapagliflozin could prevent acute graft-versus-host disease (aGVHD) in patients undergoing allogeneic hematopoietic cell transplantation (allo-HCT) with haploidentical or unrelated donor and to assess its safety. The main questions it aims to answer are: Dose Dapagliflozin lower the cumulative incidence of aGVHD? What medical problems do participants undergoing allo-HCT from haploidentical or unrelated donor have when taking Dapagliflozin? Researchers will document the occurrence of graft-versus-host disease, hematopoietic reconstitution, survival rates and adverse effects. Participants will take Dapagliflozin every day in -1 to 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65 years old.
* Patients with hematologic malignancies indicated for allo-HCT and having a suitable haploidentical or unrelated donor.
* Willing to undergo myeloablative conditioning and graft-versus-host disease prophylaxis base on cyclosporin A and methotrexate.
* With Eastern Cooperative Oncology Group (ECOG) performance status of 0-3.
* Patients with prior use of Dapagliflozin or other hypoglycemic medications may switch to Dapagliflozin, contingent upon the treating physician's assessment of contraindications, will be eligible.
* Signing an informed consent form, having the ability to comply with study and follow-up procedures.

Exclusion Criteria:

* With other malignancies.
* With a previous history of autologous hematopoietic cell transplantation, allo-HCT or chimeric antigen receptor T-cell therapy.
* With a history of allergies to Dapagliflozin.
* With type 1 diabetes or a history of ketoacidosis.
* With a history of recurrent urinary tract infections.
* With severe organ dysfunction.
* With active hepatitis B virus, hepatitis C virus, or human immunodeficiency virus infection.
* In pregnancy or lactation period.
* With any conditions not suitable for the trial (investigators' decision).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-04-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of grade II-IV aGVHD | 100 days after transplantation.
  estimated cumulative incidence of grade II-IV aGVHD at 100 days.

SECONDARY OUTCOMES:
Cumulative incidence of grade III-IV aGVHD | 100 days after transplantation.
  estimated cumulative incidence of grade III-IV aGVHD at 100 days.
Neutrophil reconstitution | up to 30 days.
  time of neutrophil reconstitution.
Platelet reconstitution | up to 100 days.
  time of platelet reconstitution.
Cumulative incidence of chronic graft-versus-host disease (cGVHD) | 1 year after transplantation.
  estimated cumulative incidence of cGVHD at 1 year.
Overall survival | 1 year after transplantation.
  estimated overall survival at 1 year.
Cumulative incidence of relapse | 1 year after transplantation.
  estimated cumulative incidence of relapse at 1 year.
Graft-versus-host disease-free relapse-free survival (GRFS) | 1 year after transplantation.
  estimated GRFS at 1 year.
Treatment related non-hematological grade 3 or higher adverse events | up to 100 days.
  Number of unique patients who had a treatment related (possible, probable or definite) non-hematological adverse event that was graded 3 or greater.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cheng Q, Wang D, Lai X, Liu Y, Zuo Y, Zhang W, Lei L, Chen J, Liu H, Wang Y, Liu H, Zheng H, Wu D, Xu Y. The OTUD1-Notch2-ICD axis orchestrates allogeneic T cell-mediated graft-versus-host disease. Blood. 2023 Mar 23;141(12):1474-1488. doi: 10.1182/blood.2022017201. PMID 36574342